CLINICAL TRIAL: NCT06069024
Title: Population Pharmacokinetic Study Based on Quantitative Pharmacology in Patients With Lenalidomide
Status: Completed | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xin Huang, Chief pharmacist, Qianfoshan Hospital
Other Study IDs: QY-SH-2021-LD-PK-001
Record Dates: First submitted 2023-09-26; First posted 2023-10-05 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma; Myelodysplastic Syndromes; Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Myelodysplastic Syndromes; Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-intervention, prospective, open-label and observational clinical trial. The researchers plan to recruit at least 50 qualified patients. The main purpose of this study was to establish a population pharmacokinetic(PPK) model of lenalidomide and explore factors associated with the adverse events of lenalidomide from a pharmacokinetic(PK) perspective.

DETAILED DESCRIPTION:
Studies have found that there is significant interpatient variability in the plasma concentration of lenalidomide, and the PK parameters of lenalidomide do not affect its efficacy but may be correlated with its toxicity. Therefore, the investigators plan to conduct a PPK study on lenalidomide to identify factors contributing to interpatient PK differences, thus refining regimens to mitigate its adverse reactions, in the hope of optimizing the clinical application of lenalidomide. At least 50 patients are planned to be included. It should be noted that the study does not interfere with the patients' treatment plans. Except for the discomfort during blood sampling, patients will not be exposed to any risks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are above the age of 18
* Patients who receive lenalidomide treatment

Exclusion Criteria:

* Patients have received other investigational systemic drugs
* The clinical data are deemed insufficient
* There appear other factors that rendered them ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with different diagnosis are eligible if they were above the age of 18 and received lenalidomide treatment.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
drug blood concentration | 2 years
  Blood samples of patients who took lenalidomide were collected by opportunistic blood collection, which were used for concentration determination by using HPLC/MS. Lenalidomide blood levels in patients were prevalent between 1-1000 ng/ml.
genotype | 1 month
  Genotypes of patients needed to be determined include ABCB1 3435 C>T, ABCB1 1236 A>G and ABCB1 2677 A>C/T.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China